CLINICAL TRIAL: NCT07167342
Title: The Effect of Oral Clostridium Butyricum on the Recurrence After Colonoscopic Resection of Colorectal Adenoma - A Multicenter, Double-blinded, Differential Design, Randomized, Placebo-controlled Study
Brief Title: The Effect of Oral Clostridium Butyricum on the Recurrence After Colonoscopic Resection of Colorectal Adenoma
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Linyi People's Hospital (Other); Shandong Cancer Hospital and Institute (Other); Yantai Yuhuangding Hospital (Other); Jining First People's Hospital (Other); Rizhao People's Hospital (Other); Qianfoshan Hospital (Other); Weifang People's Hospital (Other); Qilu Hospital of Shandong University (Other); Taian City Central Hospital (Other); The Affiliated Hospital of Shandong Second Medical University (Unknown); Dongying People's Hospital (Other)
Responsible Party: Principal Investigator, Zhou Yanbing, The Director of the Department of Gastrointestinal Surgery, the Affiliated Hospital of Qingdao University, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DHQDFY-01
Record Dates: First submitted 2025-08-26; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Adenoma; Probiotics
Keywords: Colorectal Adenoma; Clostridium butyricum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clostridium butyricum group (Experimental): Oral Clostridium butyricum capsules, Live: take 3 capsules twice daily (bid) for the first 3 months after adenoma resection, then continue with 3 capsules once daily (qd) until 3 years post-resection (each capsule contains ≥6.3 × 10⁶ CFU of Clostridium butyricum).
  Interventions: Drug: Clostridium butyricum capsules, Live
- Placebo group (Placebo Comparator): Placebo capsules containing corn starch, with identical appearance, weight, and administration method as the study group.
  Interventions: Other: Control (placebo)

INTERVENTIONS:
Drug: Clostridium butyricum capsules, Live — Oral Clostridium butyricum capsules, Live: take 3 capsules twice daily (bid) for the first 3 months after adenoma resection, then continue with 3 capsules once daily (qd) until 3 years post-resection (each capsule contains ≥6.3 × 10⁶ CFU of Clostridium butyricum).
  Arms: Clostridium butyricum group
Other: Control (placebo) — Placebo capsules containing corn starch, with identical appearance, weight, and administration method as the treatment group.
  Arms: Placebo group

SUMMARY:
The prevention of recurrence after colorectal adenoma resection remains an urgent medical issue to be addressed. Previous studies have mainly focused on nonsteroidal anti-inflammatory drugs, calcium supplements, and vitamins. The gut microbiota and its metabolic products are believed to play a potential role in the development and progression of colorectal adenomas. Clostridium butyricum, a butyrate-producing probiotic, has not yet been studied for its potential in preventing the recurrence of colorectal adenomas following resection. Therefore, this study, designed as a multicenter, double-blind, placebo-controlled randomized controlled trial, aims to explore evidence-based data on the role of Clostridium butyricum in preventing colorectal adenoma recurrence.

DETAILED DESCRIPTION:
Statistical Analysis Plan

Full Analysis Set (FAS):

Defined as all randomized subjects who received at least one dose of the assigned intervention and had at least one scheduled colonoscopy follow-up record.

Per Protocol Set (PPS):

Defined as subjects in the Clostridium butyricum group who received at least 80% of the total prescribed intervention, underwent at least two scheduled colonoscopy follow-ups, and did not use any prohibited medications specified in the protocol.

Safety Set (SS):

Defined as all subjects who received at least one dose of the intervention and had at least one safety assessment.

Primary Outcome Analysis The 3-year recurrence rate of adenomas will be analyzed using the chi-square (χ²) test.

Secondary Outcome Analysis For normally distributed continuous variables: independent-samples t-test. For skewed continuous variables and ordinal data: Mann-Whitney U test. For unordered categorical data: chi-square (χ²) test or Fisher's exact test. For repeated measures data: repeated measures ANOVA or Generalized Estimating Equations (GEE).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* No restriction on sex
* Boston Bowel Preparation Score (BBPS) ≥ 7 prior to endoscopic procedure
* Completed endoscopic resection of colorectal adenomas (including cold snare polypectomy, ESD, EMR, etc.) with no residual adenomas or polyps observed endoscopically
* Histologically confirmed adenomas (including tubular, villous, or tubulovillous types) without malignant transformation
* Able to take oral medication
* Signed informed consent

Exclusion Criteria:

* Use of probiotics, prebiotics, synbiotics, or antibiotics within 2 weeks prior to enrollment
* Presence of psychiatric disorders or other conditions preventing compliance with the intervention
* Dysfunction of vital organs (liver, kidney, heart, etc.) deemed unsuitable for clinical study participation after evaluation
* Participation in other clinical trials within 3 months prior to enrollment
* History of gastrointestinal surgery (excluding endoscopic procedures)
* History of inflammatory bowel disease
* History of autoimmune diseases
* Long-term use of aspirin (≥100 mg/day for over 3 months) or calcium supplements (≥1200 mg/day for over 3 months)
* Pregnancy or breastfeeding
* Previous treatment for colorectal adenomas (including endoscopic or surgical resection)
* Familial adenomatous polyposis (FAP)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-10-31 (Estimated); Primary Completion 2029-10-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
3-year adenoma recurrence rate | 3 years
  Each subject will undergo a colonoscopy once per year after enrollment to monitor for adenoma recurrence.
  The 3-year recurrence rate is calculated as:
  3-year recurrence rate (%) = (Number of subjects with adenoma recurrence / Total number of subjects) × 100%

SECONDARY OUTCOMES:
1-year adenoma recurrence rate | 1-year after enrollment
  Each subject will undergo a colonoscopy once per year after enrollment to monitor for adenoma recurrence.
  The 1-year recurrence rate is calculated as:
  1-year recurrence rate (%) = (Number of subjects with adenoma recurrence during the first year after enrollment/ Total number of subjects) × 100%
incidence of colorectal cancer | 3 years after enrollment
  Each subject will undergo a colonoscopy once per year after enrollment to monitor for the development of colorectal cancer.
  The incidence of colorectal cancer is calculated as:
  Incidence (%) = (Number of subjects diagnosed with colorectal cancer / Total number of subjects) × 100%
Incidence of advanced colorectal adenomas | 3 years after enrollment
  Each subject will undergo a colonoscopy once per year after enrollment to monitor for the presence of advanced adenomas.
  The incidence of advanced adenomas is calculated as:
  Incidence (%) = (Number of subjects with advanced adenomas / Total number of subjects) × 100%
  Advanced colorectal adenoma is diagnosed when any of the following criteria are met: Adenoma diameter ≥ 10 mm，Villous component ≥ 25%，Presence of high-grade intraepithelial neoplasia.
Location of adenoma recurrence | 3 years
  Classify the locations according to ascending colon, transverse colon, descending colon, sigmoid colon, and rectum.
Number of recurrent adenomas | 3 years
Histological classification of recurrent adenomas | 3 years
  Classify the locations according to Tubular adenoma, Villous adenoma, Tubulovillous adenoma, Serrated adenoma
Size of recurrent adenomas | 3 years
  Measure the maximum diameter of the adenoma in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: 淦 Zhou, Study Chair — The Affiliated Hospital of Qingdao University
Locations (1):
- the Affiliated Hospital of QIngdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No